CLINICAL TRIAL: NCT00808275
Title: Effect of Dietary Calcium on Body Weight Regulation in Adults
Brief Title: Caloric Restriction and Body Weight in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Maciej Buchowski, Research Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010590
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Overweight
Keywords: dietary calcium; weight loss
MeSH Terms: conditions — Overweight; Weight Loss | interventions — Calcium, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dairy calcium (Experimental): Diet with dairy calcium sources
  Interventions: Dietary Supplement: Dietary calcium
- Non-dairy calcium (Experimental): Diet with non-dairy calcium sources
  Interventions: Dietary Supplement: Dietary calcium

INTERVENTIONS:
Dietary Supplement: Dietary calcium — Dairy and non-dairy calcium provided as a part of diet in the amounts of 500 mg/day and 1500 mg/day. Diet contained 70% of daily caloric requirements.

SUMMARY:
The purpose of this study is to determine the role of

1. dietary calcium in fecal fat loss and the association between lactose maldigestion, dietary calcium level and source, and weight loss induced by caloric restriction.
2. caloric restriction on biomarkers of inflammation and oxidative stress

ELIGIBILITY:
Inclusion Criteria:

* 18 -65 years old
* Healthy

Exclusion Criteria:

* Body weight more than 300 lbs (body composition measurement instrument limit) diabetes
* Heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Fat in stool as a percentage of fat intake | 3 months of diet

SECONDARY OUTCOMES:
Weight change | 3 months of diet

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Buchowski, Ph.D., Principal Investigator — Vanderbilt University

REFERENCES:
- [Derived] Buchowski MS, Hongu N, Acra S, Wang L, Warolin J, Roberts LJ 2nd. Effect of modest caloric restriction on oxidative stress in women, a randomized trial. PLoS One. 2012;7(10):e47079. doi: 10.1371/journal.pone.0047079. Epub 2012 Oct 5. PMID 23071718
- [Derived] Buchowski MS, Aslam M, Dossett C, Dorminy C, Choi L, Acra S. Effect of dairy and non-dairy calcium on fecal fat excretion in lactose digester and maldigester obese adults. Int J Obes (Lond). 2010 Jan;34(1):127-35. doi: 10.1038/ijo.2009.212. Epub 2009 Oct 13. PMID 19823185